CLINICAL TRIAL: NCT05630989
Title: A Registry to Capture Patient Outcomes With KRAS G12R Altered Advanced Pancreatic Ductal Adenocarcinoma Treated With MEK Inhibitor-based Combination Therapy
Status: Recruiting | Type: Observational
Sponsor: Mandana Kamgar, MD (Other)
Responsible Party: Sponsor-Investigator, Mandana Kamgar, MD, Assistant Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Other Study IDs: PRO00045718
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; KRAS G12R mutation; Precision medicine; Retrospective Chart Review; Prospective Chart Review
MeSH Terms: interventions — Combined Modality Therapy; Hydroxychloroquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Therapy with no MEKi: Subjects have advanced PDAC with KRAS G12R mutation. Subjects' tumors must have KRAS G12R mutation, as determined by a next generation sequencing (NGS) panel or circulating tumor DNA panel of choice of the treating physician. Subjects will receive therapy with no MEKi.
  Interventions: Other: combination therapy with no MEKi
- Therapy with MEKi- Hydroxychloroquine (HCQ): Subjects have advanced PDAC with KRAS G12R mutation. Subjects' tumors must have KRAS G12R mutation, as determined by a next generation sequencing (NGS) panel or circulating tumor DNA panel of choice of the treating physician. Subjects will receive therapy with MEKi and HCQ.
  Interventions: Drug: combination therapy with MEKi-HCQ
- Therapy with MEKi- Epidermal growth factor receptor inhibitor (EGFRi): Subjects have advanced PDAC with KRAS G12R mutation. Subjects' tumors must have KRAS G12R mutation, as determined by a next generation sequencing (NGS) panel or circulating tumor DNA panel of choice of the treating physician. Subjects will receive combination therapy with MEKi and EGFRi.
  Interventions: Drug: combination therapy with MEKi-EGFRi
- Therapy with MEKi-Other: Subjects have advanced PDAC with KRAS G12R mutation. Subjects' tumors must have KRAS G12R mutation, as determined by a next generation sequencing (NGS) panel or circulating tumor DNA panel of choice of the treating physician. Subjects will receive combination therapy with MEKi and a specified drug combination.
  Interventions: Drug: combination therapy with MEKi.

INTERVENTIONS:
Other: combination therapy with no MEKi — This cohort will receive combination therapy with no MEKi.
  Other Names: mitogen-activated extracellular signal-regulated kinase inhibitor
  Groups: Therapy with no MEKi
Drug: combination therapy with MEKi-HCQ — This cohort will receive combination therapy with MEKi-HCQ.
  Other Names: mitogen-activated extracellular signal-regulated kinase inhibitor with hydroxychloroquine
  Groups: Therapy with MEKi- Hydroxychloroquine (HCQ)
Drug: combination therapy with MEKi-EGFRi — This cohort will receive combination therapy with MEKi-EGFRi.
  Other Names: mitogen-activated extracellular signal-regulated kinase inhibitor with epidermal growth factor receptor inhibitor
  Groups: Therapy with MEKi- Epidermal growth factor receptor inhibitor (EGFRi)
Drug: combination therapy with MEKi. — This cohort will receive combination therapy with MEKi.
  Other Names: mitogen-activated extracellular signal-regulated kinase inhibitor
  Groups: Therapy with MEKi-Other

SUMMARY:
This is an observational precision oncology study designed to collect and analyze data that allows us to characterize the safety and efficacy of several different mitogen-activated protein kinase kinase inhibitor (MEKi) -based treatment strategies and the feasibility of administering MEKi combination therapies to patients with KRAS G12R mutated advanced pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
Patient medical records, obtained both retrospectively and prospectively, will be examined for results of molecular profiling obtained through standard of care testing to help understand how well KRAS G12R pancreatic patients respond to MEKi-based combination matched therapy. Patient outcome parameters including but not limited to tumor response, patient survival, and toxicity will be analyzed. Moreover, metrics will be collected to ascertain whether a future clinical trial involving a MEKi-based combination therapy is feasible to carry out.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Diagnosis of advanced pancreatic ductal adenocarcinoma as determined by the treating physician or tumor board.
3. Tumor must have KRAS G12R mutation, as determined by a next generation sequencing (NGS) panel or circulating tumor DNA panel of choice of the treating physician.
4. Ability to understand a written informed consent document and the willingness to sign it.

Exclusion Criteria:

1. Age <18 years.
2. Primary cancer diagnosis other than advanced pancreatic ductal adenocarcinoma
3. Tumor does not have a KRAS G12R mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects have advanced PDAC with KRAS G12R mutation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with no progression. | 6 months
  This is defined as the time from the start of treatment until six months on treatment, or disease progression, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death, whichever occurs first.

SECONDARY OUTCOMES:
The number of subjects who have a complete response. | 2 years
  A complete response will be determined using RECIST v1.1.
The number of subjects who have a partial response. | 2 years
  A partial response will be determined using RECIST v1.1.
The number of grade 3 adverse events at least possibly related to a drug. | 2 years
  Adverse events and serious adverse events will be classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.
The number of grade 4 adverse events at least possibly related to a drug. | 2 years
  Adverse events and serious adverse events will be classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Kamgar, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No